CLINICAL TRIAL: NCT01125293
Title: Phase I/II Study of Combination Everolimus (RAD001), and Rituximab (Rituxan), OR Everolimus, Bortezomib (Velcade, PS-341), and Rituximab in Patients With Relapsed and/or Relapsed/Refractory Waldenstrom's Macroglobulinemia
Brief Title: Everolimus, Bortezomib and/or Rituximab in Patients With Relapsed/Refractory Waldenstrom's Macroglobulinemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Per protocol, Phase II is to be terminated early if a less than 5% of the Phase II participants observe a Very Good Partial Response or Better in the first 23 participants enrolled to Phase II.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry); Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Irene Ghobrial, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-280; R01FD003743; X05310 (Other Grant/Funding Number: FDAOOPD; Millennium); R01FD003743 (NIH)
Record Dates: First submitted 2010-03-16; First posted 2010-05-18 (Estimated); Results first posted 2021-04-23 (Actual); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Waldenstrom's Macroglobulinemia
Keywords: everolimus; rituximab; bortezomib; RAD001; Rituxan; Velcade
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — Everolimus; Rituximab; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase I Stage A Level 1 (Experimental): Combination of everolimus & rituximab for 6 cycles:
  Everolimus 5 mg: Taken orally on a daily basis x 28 days
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only
  (1 cycle = 28 days)
  Maintenance:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  (1 cycle = 28 days)
  Participants are treated on everolimus maintenance until progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Everolimus; Drug: Rituximab
- Phase I Stage A Level 2 (Experimental): Combination of everolimus & rituximab for 6 cycles:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only
  (1 cycle = 28 days)
  Maintenance:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  (1 cycle = 28 days)
  Participants are treated on everolimus maintenance until progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Everolimus; Drug: Rituximab
- Phase I Stage B Level 1 (Experimental): Combination of everolimus & rituximab with bortezomib for 6 cycles:
  Everolimus 5 mg: Taken orally on a daily basis x 28 days
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only
  Bortezomib 1.6 mg/m^2: Given intravenously on days 1, 8 and 15 of every cycle (1 cycle = 28 days)
  Maintenance:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  (1 cycle = 28 days)
  Participants are treated on everolimus maintenance until progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Everolimus; Drug: Rituximab; Drug: Bortezomib
- Phase I Stage B Level 2 (Experimental): Combination of everolimus & rituximab with bortezomib for 6 cycles:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only
  Bortezomib 1.6 mg/m^2: Given intravenously on days 1, 8 and 15 of every cycle
  (1 cycle = 28 days)
  Maintenance:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  (1 cycle = 28 days)
  Participants are treated on everolimus maintenance until progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Everolimus; Drug: Rituximab; Drug: Bortezomib
- Phase I Dose Expansion (Experimental): Combination of everolimus & rituximab with bortezomib for 6 cycles:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only
  Bortezomib 1.6 mg/m^2: Given intravenously on days 1, 8 and 15 of every cycle
  (1 cycle = 28 days)
  Maintenance:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  (1 cycle = 28 days)
  Participants are treated on everolimus maintenance until progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Everolimus; Drug: Rituximab; Drug: Bortezomib
- Phase II (Experimental): Combination of everolimus & rituximab with bortezomib for 6 cycles:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only
  Bortezomib 1.6 mg/m^2: Given intravenously on days 1, 8 and 15 of every cycle
  Maintenance:
  Everolimus 10 mg: Taken orally on a daily basis x 28 days
  (1 cycle = 28 days)
  Participants are treated on everolimus maintenance until progression, unacceptable toxicity or withdrawal for other reasons.
  Interventions: Drug: Everolimus; Drug: Rituximab; Drug: Bortezomib

INTERVENTIONS:
Drug: Everolimus
  Other Names: RAD001
Drug: Rituximab
  Other Names: Rituxan
Drug: Bortezomib
  Other Names: Velcade; PS-341
  Arms: Phase I Dose Expansion; Phase I Stage B Level 1; Phase I Stage B Level 2; Phase II

SUMMARY:
The purpose of this research study is to test the safety of the combination of everolimus, rituximab and bortezomib. Everolimus is a drug that works by preventing cells in your body from growing and dividing. Information from basic and other clinical research suggests that everolimus may also inhibit tumor growth in people with relapsed or refractory lymphoma. The FDA has approved everolimus for the treatment of multiple myeloma, a cancer that is closely related to Waldenstrom's Macroglobulinemia. Rituximab is approved by the FDA for the treatment of non-Hodgkin's lymphoma, which included Waldenstrom's Macroglobulinemia.

Funding Source - FDA OOPD

DETAILED DESCRIPTION:
Study Design

This is a phase I/II study. The phase I portion of the study will determine the maximum tolerated dose of everolimus, rituximab, and bortezomib combination, while the phase II portion will evaluate the depth of responses to the everolimus, rituximab, and bortezomib combination. If patients show response, they will continue on therapy for a total of 6 cycles, and then go on maintenance therapy with everolimus alone until progression. Patients on maintenance will be monitored every 3 months for response. Because of the potential of an IgM flare after rituximab, patients who show an increase in IgM after rituximab in the first 3 months will not be deemed as having progressive disease unless they show evidence of clinical progression and not just an increase of IgM levels. If biochemical progression is confirmed by m-spike, but the participant is clinically benefitting from therapy, the participant may continue on treatment for a few additional points of assessment and re-discuss benefit of therapy. Additionally, if the participant progressed because the treatment was held, participant may remain on study at the discretion of the overall Principal Investigator. Relapse from CR is defined by the reappearance of monoclonal IgM protein and/or recurrence of bone marrow involvement, lymphadenopathy/splenomegaly or symptoms attributable to active disease (Owen et al., 2012). Progression from PR is defined by ≥ 25% increase in IgM level from lowest recorded value and confirmed by a repeat assessment. The development of new signs and symptoms of disease, including Bing Neel syndrome and histological transformation, is also considered as evidence of disease progression. An absolute increase of at least 5 g/l is required to define progression when the IgM level is the only applicable criterion (Owen et al., 2012).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Patients must have received prior therapies for their WM and have relapsed or refractory WM requiring therapy. Any number of prior therapies is acceptable. Patients must not have been refractory to rituximab. The last rituximab must be at least 3 months prior to the start of treatment. Prior treatment with bortezomib and/or everolimus is permitted.
* Measurable monoclonal IgM protein in the serum OR measurable quantitative immunoglobulin M (serum IgM).
* Lymphoplasmacytic cells in the bone marrow during any previous bone marrow biopsy.
* CD20 positive disease based on any previous bone marrow immuno-histochemistry or flow cytometric analysis performed prior to enrollment.
* ECOG Performance Status 0, 1 or 2
* Laboratory values as outlined in the protocol
* Capable of swallowing intact study medication tablets
* Life expectancy of 12 weeks or greater

Exclusion Criteria:

* Uncontrolled infection
* Other active malignancies
* Cytotoxic chemotherapy 3 weeks or less, or biologic or targeted novel therapy 2 weeks or less, or corticosteroids 2 weeks or less, or radiation therapy 2 weeks or less, or any ancillary treatment considered investigation 2 weeks or less, prior to registration. Patients may be receiving chronic corticosteroids if they are being given for disorders other than WM.
* Pregnant women, nursing women, men or women of childbearing potential who are unwilling to employ adequate contraception throughout the trial and for 8 weeks after the last dose of study treatment.
* Known to be HIV positive, or Hepatitis B positive. If the status of HIV is not known and patients are not at risk, then patients will not be specifically tested for HIV. Patients will be tested for Hepatitis B at time of screening. If patients are not considered high risk and have been vaccinated at an earlier date, results of the test are not required at the time of registration. For patients that are high risk, results must be obtained prior to registration.
* Patient has Grade 2 or higher peripheral neuropathy within 14 days of enrollment
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection fo basal cell carcinoma or squamous cell carcinoma of the skin, an in situ malignancy, or low-risk prostate cancer after curative therapy.
* Severely impaired lung function
* Uncontrolled diabetes
* Liver disease such as cirrhosis, chronic active hepatitis or chronic persistent hepatitis
* Impairment of gastrointestinal function or gastrointestinal disease
* Patients with active, bleeding diathesis
* Myocardial infarction within 6 months prior to enrollment or had NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities.
* Hypersensitivity to everolimus or other rapamycins or to is excipients
* Patients who may need or are receiving live vaccines for immunization
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irene Ghobrial, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ghobrial IM, Redd R, Armand P, Banwait R, Boswell E, Chuma S, Huynh D, Sacco A, Roccaro AM, Perilla-Glen A, Noonan K, MacNabb M, Leblebjian H, Warren D, Henrick P, Castillo JJ, Richardson PG, Matous J, Weller E, Treon SP. Phase I/II trial of everolimus in combination with bortezomib and rituximab (RVR) in relapsed/refractory Waldenstrom macroglobulinemia. Leukemia. 2015 Dec;29(12):2338-46. doi: 10.1038/leu.2015.164. Epub 2015 Jul 3. PMID 26139427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled from April 2010 to July 2013.
Groups:
- Phase I Stage A Level 1: Combination of everolimus & rituximab for 6 cycles
  Everolimus 5 mg: Taken orally on a daily basis x 28 days (1 cycle)
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only (1 cycle = 28 days)
- Phase I Stage A Level 2: Combination of everolimus & rituximab for 6 cycles
  Everolimus 10 mg: Taken orally on a daily basis x 28 days (1 cycle)
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only (1 cycle = 28 days)
- Phase I Stage B Level 1: Combination of everolimus & rituximab with bortezomib for 6 cycles
  Everolimus 5 mg: Taken orally on a daily basis x 28 days (1 cycle)
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only (1 cycle = 28 days)
  Bortezomib 1.6 mg/m^2: Given intravenously on days 1, 8 and 15 of every cycle (1 cycle = 28 days)
- Phase I Stage B Level 2; Phase I Dose Expansion; Phase II: Combination of everolimus & rituximab with bortezomib for 6 cycles
  Everolimus 10 mg: Taken orally on a daily basis x 28 days (1 cycle)
  Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only (1 cycle = 28 days)
  Bortezomib 1.6 mg/m^2: Given intravenously on days 1, 8 and 15 of every cycle (1 cycle = 28 days)
Period: Overall Study
Arm/Group | Phase I Stage A Level 1 | Phase I Stage A Level 2 | Phase I Stage B Level 1 | Phase I Stage B Level 2 | Phase I Dose Expansion | Phase II
Started | 3 | 3 | 4 | 3 | 10 (Per protocol, a 10 patient expansion cohort is used to confirm the MTD determined in Stage B .) | 23
Evaluable for Phase I Dose-Limiting Toxicity | 3 | 3 | 3 | 3 | 0 (The Phase I dose expansion cohort was not evaluated for cycle 1 dose-limiting toxicity.) | 0 (The Phase II cohort was not evaluated for cycle 1 dose-limiting toxicity.)
Completed (Since treatment was not of fixed duration, all participants were considered as 'Not Completed' and reason off-treatment is provided.) | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 4 | 3 | 10 | 23
Not completed — Disease Progression | 1 | 3 | 4 | 3 | 5 | 12
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 2 | 8
Not completed — Symptomatic Deterioration | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Stage A Level 1 | Phase I Stage A Level 2 | Phase I Stage B Level 1 | Phase I Stage B Level 2 | Phase I Dose Expansion | Phase II | Total
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 10 | 23 | 46
Age, Customized [Count of Participants; unit: Participants]
  <=50 years | 0 | 0 | 0 | 1 | 0 | 3 | 4
  >50 and <=60 years | 1 | 1 | 2 | 1 | 4 | 2 | 11
  >60 and <=70 years | 2 | 1 | 2 | 1 | 5 | 12 | 23
  70+ years | 0 | 1 | 0 | 0 | 1 | 6 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2 | 2 | 3 | 11 | 20
  Male | 3 | 1 | 2 | 1 | 7 | 12 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not Hispanic or Latino | 3 | 3 | 4 | 3 | 10 | 22 | 45
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 2 | 3 | 4 | 3 | 10 | 22 | 44
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Study Site [Count of Participants; unit: Participants]
  Colorado Blood Cancer Institute | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Dana Farber Cancer Institute | 3 | 3 | 4 | 3 | 10 | 21 | 44
  Morale, Welfare, and Recreation | 0 | 0 | 0 | 0 | 0 | 1 | 1
Disease Status [Count of Participants; unit: Participants]
  Refractory | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Relapsed | 0 | 0 | 1 | 2 | 6 | 6 | 15
  Relapsed and Refractory | 0 | 0 | 0 | 0 | 0 | 3 | 3
ECOG Performance Status [Count of Participants; unit: Participants]
  00 - Fully Active | 3 | 3 | 4 | 3 | 8 | 13 | 34
  01 - Restricted | 0 | 0 | 0 | 0 | 2 | 7 | 9
  02 - Ambulatory and Capable of Self Care | 0 | 0 | 0 | 0 | 0 | 3 | 3
International Prognostic Scoring System for Waldenstrom Macroglobulinemia [Count of Participants; unit: Participants] — Low is defined as 1 or dewer of the following:
  Hemoglobin (HB) <=11.5 g/dL Platelet (PT) <=100 x 10^9 / L Beta 2 Microglubin (B2M) > 3 mg/L Immunoglobulin M (IgM) > 7 g/dL
  Intermediate is defined as over 65 years old or two of the following:
  HB <=11.5 g/dL PT <=100 x 10^9 / L B2M > 3 mg/L IgM> 7 g/dL
  High is defined as more than 2 of the following:
  Over 65 years old HB <=11.5 g/dL PT <=100 x 10^9 / L B2M > 3 mg/L IgM> 7 g/dL
  Participants
    Low | 2 | 1 | 1 | 2 | 6 | 6 | 18
    Intermediate | 0 | 1 | 2 | 1 | 4 | 13 | 21
    High | 1 | 1 | 1 | 0 | 0 | 4 | 7
Number of Prior Therapies (Continuous) [Median (Full Range); unit: number of therapies] | 5 [2 to 6] | 3 [1 to 4] | 2 [2 to 8] | 1 [1 to 2] | 2 [1 to 7] | 2 [1 to 9] | 2 [1 to 9]
Prior Rituximab Treatment [Count of Participants; unit: Participants]
  No | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Yes | 3 | 3 | 4 | 3 | 10 | 22 | 45
Prior Bortezomib Treatment [Count of Participants; unit: Participants]
  No | 0 | 2 | 2 | 1 | 5 | 10 | 20
  Yes | 3 | 1 | 2 | 2 | 5 | 13 | 26
Prior Rituximab/Bortezomib Combination Treatment [Count of Participants; unit: Participants]
  No | 0 | 2 | 2 | 1 | 5 | 11 | 21
  Yes | 3 | 1 | 2 | 2 | 5 | 12 | 25
Time from Initial Diagnosis to Study Entry (Months) [Median (Full Range); unit: month] — Population: One participant in the Dose Expansion arm had missing data for this measure.
  month
    number analyzed (Participants) | 3 | 3 | 4 | 3 | 10 | 22 | 45
    (all) | 142.2 [38.3 to 170.4] | 83.9 [16.7 to 131.8] | 61.8 [57.0 to 115.2] | 38.2 [4.9 to 70.7] | 48.2 [16.2 to 163.2] | 64.5 [5.3 to 250.7] | 63.1 [4.9 to 250.7]

OUTCOME MEASURES:

1. Primary Outcome: Everolimus Maximum Tolerated Dose (MTD) Stage A [Phase I]
Description: The MTD of Everolimus/Rituximab combination is determined by the number of patients who have dose limiting toxicity (DLT). See DLT primary outcome measure for definition. MTD is defined as the highest dose where <1/3 participants experience a DLT. If no DLT's are observed on Level 1, 3 subjects will be enrolled in the Level 2. If >1/3 subjects in a cohort have DLT, that dose will not be considered safe, with no escalation (MTD exceeded). If 1/3 subjects experience DLT, the cohort will be expanded to 6 subjects. If <2 subjects with a DLT among the expanded cohort of 6 evaluable subjects a cohort of 3 subjects will be enrolled in the next higher dose level. If 2 or more subjects with a DLT among the expanded cohort of 6 subjects, that dose level will not be considered safe, no escalation (MTD exceeded). If no DLT's are observed, then the MTD is not reached. The MTD was not reached with 0/3 participants experiencing a DLT in the highest dose level. Higher doses were not planned/tested.
Time Frame: Assessed within the first cycle (28 days) of the study.
Population: The analysis dataset includes all participants enrolled to Stage A.
Measure: Number; unit: mg
Groups:
- Phase I Stage A Level 1 and 2: Combination of everolimus & rituximab for 6 cycles:
  Level 1:Everolimus 5 mg: Taken orally on a daily basis x 28 days (1 cycle)
  Level 2:Everolimus 10 mg: Taken orally on a daily basis x 28 days (1 cycle)
  Levels 1 and 2: Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only (1 cycle = 28 days)
Arm/Group | Phase I Stage A Level 1 and 2
Number analyzed (Participants) | 6
mg | 10

2. Primary Outcome: Everolimus Maximum Tolerated Dose (MTD) Stage B [Phase I]
Description: The MTD of Everolimus/Bortezomib/Rituximab combination is determined by the number of patients who have dose limiting toxicity (DLT). See DLT primary outcome measure for definition. MTD is defined as the highest dose where <1/3 participants experience a DLT. If no DLT's are observed on Level 1, 3 subjects will be enrolled in the Level 2. If >1/3 subjects in a cohort have DLT, that dose will not be considered safe, with no escalation (MTD exceeded). If 1/3 subjects experience DLT, the cohort will be expanded to 6 subjects. If <2 subjects with a DLT among the expanded cohort of 6 evaluable subjects a cohort of 3 subjects will be enrolled in the next higher dose level. If 2 or more subjects with a DLT among the expanded cohort of 6 subjects, that dose level will not be considered safe, no escalation (MTD exceeded).If no DLT's observed, then the MTD is not reached. The MTD was not reached with 0/3 participants experiencing a DLT in the highest level. Higher doses were not planned/tested.
Time Frame: Assessed within the first cycle (28 days) of the study.
Population: In Phase I Stage B Level 1, one participant was replaced as an exception granted to the principal investigator having experienced a dose delay due to an adverse event not deemed a DLT.
Measure: Number; unit: mg
Groups:
- Phase I Stage B Level 1 & 2 and Dose Expansion: Combination of everolimus & rituximab with bortezomib for 6 cycles
  Level 1: Everolimus 5 mg: Taken orally on a daily basis x 28 days (1 cycle)
  Level 2 and Dose Expansion: Everolimus 10 mg: Taken orally on a daily basis x 28 days (1 cycle)
  Level 1 & 2 and Dose Expansion: Rituximab 375 mg/Kg: Given intravenously on days 1, 8, 15 and 22 of Cycle 1 and Cycle 4 only (1 cycle = 28 days)
  Level 1 & 2 and Dose Expansion: Bortezomib 1.6 mg/m^2: Given intravenously on days 1, 8 and 15 of every cycle (1 cycle = 28 days)
Arm/Group | Phase I Stage B Level 1 & 2 and Dose Expansion
Number analyzed (Participants) | 6
mg | 10

3. Primary Outcome: Everolimus Dose Limiting Toxicity (DLT) [Phase I]
Description: The following qualify as dose limiting toxicities:
  * Grade 3 or greater non-hematologic toxicity, considered by the investigator to be related to study drugs.
  * Grade 4 hematologic toxicity defined as: thrombocytopenia with platelets <10,000 µ/L on more than one occasion despite transfusion support; grade 4 neutropenia occurring for more than 7 days and/or resulting in neutropenic fever with elevated temperature (defined as > 101 degrees F). Lymphopenia, a recognized side effect of bortezomib, is not considered a DLT.
  * Inability to receive Day 1 dose for Cycle 2 due to toxicity
Time Frame: Assessed within the first cycle (28 days) of the study.
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Phase I Stage A Level 1 | Phase I Stage A Level 2 | Phase I Stage B Level 1 | Phase I Stage B Level 2
Number analyzed (Participants) | 3 | 3 | 3 | 3
participants | 0 | 0 | 0 | 0

4. Primary Outcome: Very-good-partial-response-or-better Rate [Phase II]
Description: Very-good-partial-response-or-better rate is the percentage of participants with complete response (CR) or very good partial response (VGPR) on to the combination of everolimus/bortezomib/rituximab. The combination regimen was received for up to 6 cycles.
  CR:
  * Absence of serum monoclonal IgM protein by immunofixation
  * Normal serum IgM level
  * Complete resolution of extramedullary disease, i.e., lymphadenopathy and splenomegaly if present at baseline
  * Morphologically normal bone marrow aspirate and trephine biopsy
  VGPR:
  * Monoclonal IgM protein is detectable ≥90% reduction in serum IgM level from baseline*
  * Complete resolution of extramedullary disease, i.e.
Time Frame: Up to 6 cycles (Day 168)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 23
percentage of participants | 4.3 [0 to 19]
Statistical Analysis 1: Comparison: Phase II; In a two-stage Simon design, a VGPR or better rate of at least 18% is considered promising versus a 5% or less rate. In stage 1, if 1 or fewer of 23 evaluable participants achieve VGPR, the regimen is considered non-promising else continue with 24 more patients enrolled. If </=4 of 47 evaluable patients have VGPR or better, the regimen is considered non-promising. If >/=5, then the regimen is considered promising for further study. With this design, there is 90% power and 1-sided 10% alpha; Test type: Other; p = 0.69, Two stage design, exact method; The study did not continue to stage 2 given 1 VGPR or better response was observed in 23 evaluable participants in stage 1

5. Secondary Outcome: Treatment-Emergent Sensory Neuropathy Rate [Phase I]
Description: Percentage of participants experiencing Grade 1 - Grade 3 treatment-emergent peripheral (sensory) neuropathy events based on CTCAEv3 as reported on case report forms for phase I participants.
Time Frame: Adverse events were assessed each cycle (ever 28 days) for 6 cycles then every 3 months on maintenance. Duration of therapy for the Phase I study up to 41 months.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase I Stage A Level 1 | Phase I Stage A Level 2 | Phase I Stage B Level 1 | Phase I Stage B Level 2 | Phase I Dose Expansion | Phase II
Number analyzed (Participants) | 3 | 3 | 4 | 3 | 10 | 23
percentage of participants | 33 [6 to 80] | 33 [6 to 80] | 100 [51 to 100] | 67 [21 to 94] | 50 [24 to 76] | 48 [29 to 67]

6. Secondary Outcome: Phase II Overall Response Rate
Description: Overall response rate is percentage of participants with complete (CR), very good partial (VGPR), partial (PR), or minimal response (MR) as best response during treatment.
  CR:
  * No serum monoclonal IgM protein by immunofixation
  * Normal IgM level
  * Complete resolution of extramedullary disease, i.e., lymphadenopathy and splenomegaly if present at baseline
  * Morphologically normal bone marrow aspirate and trephine biopsy
  VGPR:
  * Monoclonal IgM protein is detectable ≥90% reduction in IgM level from baseline
  * Complete resolution of extramedullary disease, i.e., lymphadenopathy/splenomegaly if present at baseline
  * No new signs/symptoms of active disease
  PR:
  * Monoclonal IgM protein is detectable ≥50% but <90% reduction in IgM level from baseline
  * Reduction in extramedullary disease
  * No new signs/symptoms of active disease
  MR:
  * Monoclonal IgM protein is detectable ≥25% but <50% reduction in IgM level from baseline
  * No new signs/symptoms of active disease
Time Frame: Up to 6 cycles (Day 168)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 23
percentage of participants | 87 [70 to 96]

7. Secondary Outcome: 2-year Time-to-progression Probability (TTP) [Phase II]
Description: 2-year TTP probability is based on Kaplan-Meier methods. TTP is defined as time from enrollment to the date of progressive disease (PD). PD is defined as ≥25% increase in serum IgM level from lowest nadir and/or progression in clinical features attributable the disease. Patients without PD and not reporting use of non-protocol therapy prior to PD are censored at date of last objective progression-free disease assessment. Patients reporting use of non-protocol therapy prior to PD are censored at date of last objective progression-free disease assessment date prior to post-discontinuation therapy.
Time Frame: Patients were assessed for disease every cycle while on treatment (168 days) and every three months while on maintenance therapy. In long-term follow-up, disease was monitored every 3 months. Study cohort median (range) follow-up was 15 (1 - 23) months.
Measure: Number (95% Confidence Interval); unit: percent probability of progression
Arm/Group | Phase II
Number analyzed (Participants) | 23
percent probability of progression | 28 [5 to 57]

8. Secondary Outcome: 2 Year Progression-free-survival [Phase II]
Description: 2-year progression free survival (PFS) is the probability of participants alive and progression free at 2 years from study entry estimated using Kaplan-Meier methods. PFS is defined as the time from enrollment to progressive disease (PD) or death. PD is defined as ≥25% increase in serum IgM level from lowest nadir and/or progression in clinical features attributable the disease. Patients alive without PD and not reporting use of non-protocol therapy prior to PD are censored at date of last objective progression-free disease assessment. Patients reporting use of non-protocol therapy prior to PD are censored at date of last objective progression-free disease assessment date prior to post-discontinuation therapy.
Time Frame: as for outcome 7
Measure: Number (95% Confidence Interval); unit: percent probability of PFS
Arm/Group | Phase II
Number analyzed (Participants) | 23
percent probability of PFS | 28 [5 to 57]

9. Secondary Outcome: Phase II Duration of Response (DoR)
Description: The DoR is defined as the elapsed time from date when the measurement criteria are first met for a complete or partial response (whichever status is recorded first) until the date of first observation of objective disease progression. Analysis of DoR will be as follows:
  * For responding patients who die without objective PD (including death from study disease), DoR will be censored at the date of the last objective progression-free disease assessment.
  * For responding patients not known to have died as of the data cut-off date and who do not have objective PD, DoR will be censored at the date of the last objective progression-free disease assessment.
  * For responding patients who receive subsequent systemic anticancer therapy (after discontinuation from the study chemotherapy) prior to objectively determined disease progression, DoR will be censored at the date of the last objective progression-free disease assessment prior to post discontinuation therapy.
Time Frame: as for outcome 7
Measure: Median (Full Range); unit: months
Arm/Group | Phase II
Number analyzed (Participants) | 23
months | 14 [1 to 23]

10. Secondary Outcome: PTEN Mutation Rate [Phase II]
Description: The PTEN mutation rate is the percentage of patients with PTEN mutation identified in pre-therapy and post-therapy bone marrow samples per established methods.
Time Frame: Samples were collected pre-therapy before the beginning therapy (baseline) and post-therapy after finishing the 6th treatment cycle (168 days).
Population: The correlative objective for the study was to identify molecular regulators of response/resistance. Because the study terminated early with limited efficacy shown in the stage 1 cohort correlative objectives could not be met. Bone marrow and peripheral blood samples were collected pre- and post-therapy for phase II patients but only a few experiments conducted considering resources and the limited potential interpretation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase II
Number analyzed (Participants) | 20
percentage of participants
  MYD88/L265P mutation | 80 [56 to 94]
  CXCR4/C1013G mutation | 5 [0 to 25]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were assessed each cycle (ever 28 days) for 6 cycles then every 3 months on maintenance therapy. In this study cohort, AE assessment was a median (range) of 10 (1-42 months).
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Phase I Stage A Level 1 | Phase I Stage A Level 2 | Phase I Stage B Level 1 | Phase I Stage B Level 2 | Phase I Dose Expansion | Phase II
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/4 | 0/3 | 1/10 | 0/23
Serious Adverse Events (participants affected / at risk) | 1/3 | 3/3 | 3/4 | 3/3 | 8/10 | 11/23
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 3/3 | 10/10 | 23/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Stage A Level 1 (N=3) | Phase I Stage A Level 2 (N=3) | Phase I Stage B Level 1 (N=4) | Phase I Stage B Level 2 (N=3) | Phase I Dose Expansion (N=10) | Phase II (N=23)
Hemoglobin (Blood and lymphatic system disorders) | 1 | 1 | 1 | 1 | 2 | 5
Infection Gr0-2 neut, lung (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection Gr0-2 neut, upper airway (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection w/ gr3-4 neut, upper airway (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection w/ unk ANC lung (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
ALT, SGPT (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Leukocytes (Investigations) | 1 | 2 | 1 | 2 | 4 | 2
Lymphopenia (Investigations) | 0 | 1 | 0 | 1 | 1 | 0
Neutrophils (Investigations) | 1 | 2 | 2 | 2 | 3 | 2
Platelets (Investigations) | 1 | 0 | 1 | 1 | 1 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy-sensory (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 1 | 0
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Skin-other (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I Stage A Level 1 (N=3) | Phase I Stage A Level 2 (N=3) | Phase I Stage B Level 1 (N=4) | Phase I Stage B Level 2 (N=3) | Phase I Dose Expansion (N=10) | Phase II (N=23)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hematologic-other (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hemoglobin (Blood and lymphatic system disorders) | 2 | 3 | 2 | 2 | 5 | 9
Lymph node, pain (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cardiac-other (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Left ventricular diastolic dysfunction (Cardiac disorders) | 0 | 0 | 0 | 0 | 2 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 3
Hearing w/w-o audiogr in monitor prg (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 2
Eyelid dysfunction (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Vision-blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdomen, pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 3
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 0 | 2 | 2 | 2 | 4 | 10
Distention/bloating, abdominal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Esophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
GI-other (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Incontinence, anal (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 2
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 0 | 1 | 3 | 3 | 3 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 2 | 1 | 2 | 3
Obstruction, small bowel NOS (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oral cavity, hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oral cavity, pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oral gums, pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Perforation, cecum (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Perforation, rectum (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rectum, pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Stomach, pain (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 2
Chest/thoracic pain NOS (General disorders) | 0 | 0 | 1 | 0 | 2 | 2
Constitutional, other (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Edema head and neck (General disorders) | 0 | 0 | 0 | 0 | 0 | 2
Edema limb (General disorders) | 0 | 0 | 2 | 1 | 2 | 8
Edema visceral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Extremity-lower (gait/walking) (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 3 | 3 | 3 | 3 | 9 | 8
Fever w/o neutropenia (General disorders) | 1 | 2 | 0 | 1 | 3 | 3
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain-other (General disorders) | 0 | 0 | 0 | 1 | 1 | 2
Rigors/chills (General disorders) | 1 | 0 | 1 | 1 | 0 | 2
Allergic reaction (Immune system disorders) | 0 | 0 | 0 | 0 | 3 | 6
Infection Gr0-2 neut, colon (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Infection Gr0-2 neut, eye NOS (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 0
Infection Gr0-2 neut, heart (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection Gr0-2 neut, lung (Infections and infestations) | 0 | 1 | 1 | 0 | 2 | 1
Infection Gr0-2 neut, middle ear (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1
Infection Gr0-2 neut, nerve-cranial (Infections and infestations) | 0 | 0 | 0 | 0 | 2 | 0
Infection Gr0-2 neut, nerve-periph (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection Gr0-2 neut, nose (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection Gr0-2 neut, salivary (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Infection Gr0-2 neut, sinus (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Infection Gr0-2 neut, stomach (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infection Gr0-2 neut, ungual (Infections and infestations) | 0 | 2 | 2 | 2 | 1 | 2
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 0 | 1 | 0 | 0 | 2 | 2
Infection w/ unk ANC bronchus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Infection w/ unk ANC lung (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 2
Infection w/ unk ANC sinus (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 3
Infection w/ unk ANC skin (cellulitis) (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 2
Infection w/ unk ANC upper airway NOS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 4
Infection w/ unk ANC urinary tract NOS (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 1
Infection-other (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Intra-op injury Heart (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 2
Alkaline phosphatase (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
AST, SGOT (Investigations) | 0 | 0 | 1 | 2 | 3 | 0
Creatinine (Investigations) | 0 | 0 | 0 | 0 | 2 | 2
Hypercholesterolemia (Investigations) | 0 | 0 | 0 | 0 | 1 | 8
Leukocytes (Investigations) | 1 | 2 | 1 | 3 | 4 | 9
Lymphopenia (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Neutrophils (Investigations) | 1 | 2 | 2 | 3 | 4 | 9
Platelets (Investigations) | 0 | 0 | 1 | 1 | 2 | 4
Weight loss (Investigations) | 0 | 0 | 0 | 1 | 0 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 5 | 8
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 2 | 9
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 1
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 9
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Back, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 2
Chest wall, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 0 | 3 | 2
Joint-function (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Muscle, pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal/soft tissue-other (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neck, pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nonneuropathic generalized weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Nonneuropathic lower extr muscle weak (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Head/headache (Nervous system disorders) | 2 | 1 | 2 | 3 | 1 | 1
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neurologic-other (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Neuropathy CN VII face-motor / taste (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Neuropathy CN VIII hearing + balance (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Neuropathy-motor (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 1
Neuropathy-sensory (Nervous system disorders) | 1 | 0 | 2 | 1 | 6 | 7
Sinus, pain (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 0
Taste disturbance (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 7
Anxiety (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 2
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bladder spasms (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 2 | 0
Incontinence urinary (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Obstruction-ureteral (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Renal/GU-other (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 2
Urinary hemorrhage NOS (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Irregular menses (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pelvic, pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 2
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 2 | 3 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 1 | 6 | 4
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 3
Pleural effusion (non-malignant) (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 2 | 1 | 5 | 7
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Throat/pharynx/larynx, pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Nail changes (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus/itching (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 4 | 2
Rash/desquamation (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 2 | 6
Sweating (Skin and subcutaneous tissue disorders) | 1 | 1 | 1 | 0 | 1 | 0
Ulceration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0
Thrombosis/thrombus/embolism (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vascular access,Thrombosis/embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes